CLINICAL TRIAL: NCT05331599
Title: Recurrence Markers, Cognitive Burden and Neurobiological Homeostasis in Late-Life Depression
Acronym: REMBRANDT
Status: Active, not recruiting | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Pittsburgh (Other); Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Olusola Alade Ajilore, Associate Professor; Associate Director, Residency Training and Education; Director, Psychiatry Residency Neuroscience Research Tracks Affiliation: University of Illinois at Chicago, University of Illinois at Chicago
Other Study IDs: 2020-0078; 1R01MH121384-01 (NIH)
Record Dates: First submitted 2020-04-08; First posted 2022-04-15 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Depression in Old Age; Recurrence; Cognitive Dysfunction
Keywords: Depression in Old Age; Recurrence; Antidepressive Agents; Depression; Neurobiological Markers; Cognitive Dysfunction; Anxiety Depression
MeSH Terms: conditions — Recurrence; Cognitive Dysfunction; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Currently Depressed Participants: Individuals who are currently depressed and receive treatment through an antidepressant treatment
- Remitted Depressed Participants: Individuals who have achieved remission from depression within 4 months
- Remitted Depressed Elders: Individuals who no lifetime history of depression

SUMMARY:
Late-life depression (LLD) is associated with disability, increased risk for cognitive decline and dementia, elevated suicide risk, and greater all-cause mortality. These outcomes are related to depression being a recurrent disorder, with repeated episodes over a patient's lifetime. Recurrence rates (defined as including both relapse and recurrence) are high in LLD.

The goals of this study are to identify neurobiological factors that predict recurrence risk, and examine how cognitive performance changes are both influenced by these neurobiological factors and also predict recurrence risk.

ELIGIBILITY:
Inclusion Criteria:

* Currently depressed participants (who will enter the treatment algorithm): 1) Age > 60 years; 2) diagnosis of major depressive disorder, recurrent episode (DSM5); 3) severity: Montgomery Asberg Depression Rating Scale (MADRS) (67) ≥ 15; 4) cognition: Montreal Cognitive Assessment (MoCA) >24 or Montreal Cognitive Assessment (MoCA) - BLIND ≥ 18; 5) fluent in English.
* Remitted depressed participants (who will directly enter the longitudinal study): 1) Age > 60 years; 2) diagnosis of major depressive disorder, recurrent, in partial or full remission (DSM5); 3) severity: MADRS < 10; 4) cognition: MoCA >24 or Montreal Cognitive Assessment (MoCA) - BLIND ≥ 18; 5) fluent in English.
* Never- depressed elders: 1) Age > 60 years; 2) severity: MADRS < 8; 3) cognition: MoCA >24 or MoCA - BLIND ≥ 18; 4) fluent in English.

Exclusion Criteria:

* Currently depressed participants (who will enter the treatment algorithm): 1) Other Axis I psychiatric disorders, except for simple phobia or anxiety disorders present during the depressive episode (e.g., generalized anxiety disorder (GAD) or panic disorder symptoms); 2) History of alcohol or drug dependence or abuse (other than nicotine) in the last year; 3) History of a developmental disorder or history of IQ < 70; 4) Acute suicidality within 3 months of study entry; 5) Acute grief (<1 month); 6) Current or past psychosis; 7) Primary neurological disorder, including dementia, clinical stroke, brain tumor, epilepsy, etc.; 8) Presence of unstable medical illness requiring urgent treatment; 9) Any MRI contraindication; 10) ECT in last 6 months; 11) Vagal Nerve Stimulation within 6 months of study entry; 12) Current use of TMS, ketamine, or esketamine with plans to continue treatment.
* Remitted depressed participants (who will directly enter the longitudinal study): Identical to the currently depressed participants, plus 1) currently receiving brain stimulation treatment (ECT, TMS, VNS), ketamine or esketamine. There are no other exclusions for antidepressant treatment.
* Never- depressed elders: Identical to the currently depressed participants, plus: 1) No diagnosis of current or past depressive disorder or other Axis I disorder except for simple phobia; 2) No history of psychotropic medication use for psychiatric symptoms.

We will not be enrolling vulnerable populations, specifically pregnant women, children, prisoners, or institutionalized individuals. We also will not enroll subjects incapable of providing their own consent. Should a potential subject present where there is a concern (either by a study clinician or staff member) about their ability to understand study procedures and provide meaningful consent, their cognitive ability and understanding will be evaluated by a study doctor. If there is any concern that the individual may be impaired, they will not be enrolled in the study. The rationale will be provided to the individual as well as his or her family members. Referrals for further evaluation, including urgent or emergent evaluation, will be made as needed and clinically warranted.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will enroll patients from clinical referrals and response to advertisements. For clinical referrals, referring providers may either provide information about the study to the participant, including our contact information. Alternatively, they may obtain permission from the participant for the study team to contact them. With the clinician's agreement, study staff can review their clinic schedules to help identify potentially eligible patients, however data will not be recorded for research purposes. Advertisements may include radio, newspapers, internet, online research registries, public transportation, and flyers / brochures.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Neurobiology of Recurrence (Stress Reactivity) | Change in stress reactivity at Month 8, Month 16, and Month 24
  Stress reactivity measured experimentally (neural reactivity during fMRI stress induction task) and ecologically (affective instability by ecological momentary assessment).
Neurobiology of Recurrence (Functional Network Connectivity) | Change in functional network connectivity at Month 8, Month 16, and Month 24
  Alterations in functional network connectivity which includes both intra/internetwork connectivity markers and well as markers of network instability.

SECONDARY OUTCOMES:
Change in Cognitive Function | Change in cognitive function at Month 0 and Month 24
  Cognition will be assessed a conventional, broad-based battery.

CONTACTS AND LOCATIONS:
Overall Officials: Amruta Barve, MPH, Study Chair — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No